CLINICAL TRIAL: NCT00278993
Title: A Phase II, Multicenter, Open Label, Two Stage Design Study Evaluating E7389 in Patients With Hormone Refractory Prostate Cancer With Advanced and/or Metastatic Disease Stratified by Prior Chemotherapy
Brief Title: Evaluating E7389 in Patients With Hormone Refractory Prostate Cancer With Advanced and/or Metastatic Disease Stratified by Prior Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-G000-204; 2005-004271-37 (EudraCT Number)
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Results first posted 2012-05-15 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2012-04

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; metastatic disease
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — eribulin

ARMS (1):
- 1 (Active Comparator): With stratification
  Interventions: Drug: E7389

INTERVENTIONS:
Drug: E7389 — Intravenous 1.4 mg/m2 on a 3-week course.

SUMMARY:
This is a multi-centre, phase II, open-label, two-stage design, single-arm study in patients with hormone-refractory prostate cancer (HRPC) with advanced (rising PSA) and/or metastatic disease and who have had prior anti-androgen therapy. The study will further explore the efficacy of E7389 by enrollment of patients into two strata: those who have had no prior systemic chemotherapy for their disease (except for mitoxantrone and estramustine), and those who failed no more than one previous chemotherapeutic regimen with tubulin-binding agents such as docetaxel.

ELIGIBILITY:
Inclusion criteria:

1. Males with histologically proven adenocarcinoma of the prostate that has progressed (ie. a minimum of 3 consecutive rises in Prostate Specific Antigen (PSA) (with the last value ≥ 4 ng/mL) taken at least 1 week apart prior to study entry) despite castration or maintenance of castrate-level testosterone (defined as serum testosterone ≤ .50 ng/dL or 1.7 nmol/L), or progressed during non-hormonal chemotherapy.

   Note: Patients previously treated with an antiandrogen must have disease progression documented after antiandrogen withdrawal. Those who have not undergone orchiectomy must continue medical castration with a gonadotropin-releasing hormone analog. At least 4 weeks must have elapsed between the withdrawal of antiandrogens (6 weeks in the case of nilutamide or bicalutamide and four weeks in the case of flutamide or other secondary hormonal therapy) and enrollment, so as to avoid the possibility of confounding results of the response due to antiandrogen withdrawal.
2. Patients must fulfill one of the following two criteria to be stratified:

   * No prior chemotherapy (except mitoxantrone or estramustine) for advanced and/or metastatic disease as defined in inclusion criteria #1.
   * Failure of no more than one previous chemotherapeutic regimen with tubulin binding agents such as docetaxel.
3. Resolution of all chemotherapy or radiation-related toxicities to less than grade 2 severity, except neuropathy and alopecia
4. Age ≥ 18 years.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2.
6. Life expectancy of ≥ 3 months.
7. Adequate renal function as evidenced by serum creatinine ≤ 1.5 times upper limits of normal (ULN) or calculated creatinine clearance ≥ 40 mL/minute (min) per the Cockcroft and Gault formula.
8. Adequate bone marrow function as evidenced by absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, hemoglobin ≥ 9.0 g/dL (or 5.5 mmol/L), and platelet count ≥ 100 x 10^9/L. Adequate liver function as evidenced by bilirubin ≤ 1.5 x ULN, alanine transaminase (ALT), and aspartate transaminase (AST) ≤ 3 x ULN (in the case of liver metastases ≤ 5 x ULN).
9. Patients willing and able to complete the VAS (Visual Analog Scale).
10. Patients willing and able to comply with the study protocol for the duration of the study.
11. Written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice.

Exclusion criteria:

1. Patients who have received chemotherapy, radiation, or experimental therapy within 4 weeks of start of E7389 treatment
2. Radiation therapy encompassing ≥30% of marrow or treatment with radioactive strontium
3. Patients who require therapeutic anti-coagulant therapy with warfarin or related compounds; (mini dose warfarin or related compounds are permitted).
4. Severe / uncontrolled intercurrent illness/infection.
5. Significant cardiovascular impairment (history of congestive heart failure > NYHA grade II, unstable angina or myocardial infarction within the past six months, or serious cardiac arrhythmia)
6. Patients with organ allografts.
7. Patients with known immunosuppression such as positive HIV status.
8. Patients who have had a prior malignancy, other than nonmelanoma skin cancer, unless the prior malignancy was diagnosed and definitively treated ≥ 5 years previously with no subsequent evidence of recurrence.
9. Patients with pre-existing neuropathy > Grade 2
10. Patients with brain or subdural metastases are not eligible, except if they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least two weeks before starting treatment with E7389.
11. Patients with meningeal carcinomatosis.
12. Patients with a hypersensitivity to halichondrin B and/or halichondrin B chemical derivative.
13. Patients who participated in a prior E7389 clinical trial.
14. Patients with other significant disease or disorders that, in the Investigator's opinion, would exclude the patient from the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2006-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asha Das, Study Director — Eisai Inc.
Locations (18):
- United States (18):
  - Dr. Robert Jotte, Denver, Colorado
  - Melbourne Internal Medicine Associates, Melbourne, Florida
  - Ocala Oncology Center PL, Ocala, Florida
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Minnesota Hematology Oncology, Burnsville, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - New York Oncology Hematology, P.C., Albany, New York
  - St. Luke's Roosevelt Hospital Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Raleigh Hematology Oncology Associates PL, Raleigh, North Carolina
  - US Oncology, Dallas, Texas
  - Mary Crowley Medical Research Center, Dallas, Texas
  - El Paso Cancer Treatment Center, El Paso, Texas
  - Texas Oncology PA, Fort Worth, Texas
  - Texas Oncology PA, Tyler, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Deke Slayton Cancer Center, Webster, Texas
  - Virginia Oncology Associates, Norfolk, Virginia

REFERENCES:
- [Derived] de Liano AG, Reig O, Mellado B, Martin C, Rull EU, Maroto JP. Prognostic and predictive value of plasma testosterone levels in patients receiving first-line chemotherapy for metastatic castrate-resistant prostate cancer. Br J Cancer. 2014 Apr 29;110(9):2201-8. doi: 10.1038/bjc.2014.189. Epub 2014 Apr 10. PMID 24722180

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 22 centers in U.S, UK, Spain and Hungary during the period of Feb 2006 to May 2009.
Groups:
- E7389 Intravenous 1.4 mg/m2: E7389 intravenous 1.4 mg/m2 on a 3-week course
Period: Overall Study
Arm/Group | E7389 Intravenous 1.4 mg/m2
Started | 108
Completed | 1
Not Completed | 107
Not completed — Adverse Event | 24
Not completed — Withdrawal by Subject | 5
Not completed — Progressive Disease | 65
Not completed — Physician Decision | 9
Not completed — Not Otherwise Specified | 4

BASELINE CHARACTERISTICS:
Arm/Group | E7389 Intravenous 1.4 mg/m2
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: years] — Intent to Treat/Safety Population
  years | 71.0 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 108
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 94
  More than one race | 0
  Other | 5
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Prostate Specific Antigen (PSA) Response Rate Based on Bubley Criteria
Description: Bubley Criteria: Patients must have progressive disease to enter study. For outcomes, PSA response must show at least 50% decrease. Duration of response is the time from >50% decrease from baseline to when there is a 50% decrease in nadir. PSA progressive disease- 25% increase from baseline or increase of 5 ng/mL along with measureable disease Stable disease- decline of less than 50% and not more than 25% increase.
Time Frame: 12 months
Population: Per Protocol Population
Measure: Number; unit: Percentage of Participants
Arm/Group | E7389 Intravenous 1.4 mg/m2
Number analyzed (Participants) | 105
Percentage of Participants
  Response | 16.2
  Stable Disease | 52.4
  Progressive Disease | 29.5
  Unknown/Not Evaluated | 1.9

2. Secondary Outcome: Duration of Prostate Specific Antigen Response Based on Bubley Criteria
Description: Duration of response is the time from >50% decrease from baseline to when there is a 50% decrease in nadir.
Time Frame: 12 months.
Population: Per Protocol Population
Measure: Median (Full Range); unit: Days
Arm/Group | E7389 Intravenous 1.4 mg/m2
Number analyzed (Participants) | 105
Days | 96 [31 to 938]

3. Secondary Outcome: Progression Free Survival
Description: From the date study treatment was initiated until the earliest date of the first PSA assessment that determined progressive disease, or the death of death if death occurred without disease progression.
Time Frame: 12 months
Population: Per Protocol Population
Measure: Median (Full Range); unit: Days
Arm/Group | E7389 Intravenous 1.4 mg/m2
Number analyzed (Participants) | 105
Days | 64 [1 to 979]

4. Secondary Outcome: Overall Survival
Time Frame: 12 months
Population: Intent to Treat Population
Measure: Median (Full Range); unit: Days
Arm/Group | E7389 Intravenous 1.4 mg/m2
Number analyzed (Participants) | 108
Days | 567 [426 to 759]

5. Secondary Outcome: Best Objective Tumor Response Rate Based on Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Based on Response Evaluation Criteria in Solid Tumors (RECIST), consisting of complete response (CR) plus partial response (PR). Defined as the best response from the start of treatment until disease progression or recurrence. Lesions measured by computed tomography (CT) scan and magnetic resonance imaging (MRI). Objective response rate: complete response (CR-disappearance of all lesions)+ partial response (PR-30% decrease in lesion diameter), Progressive Disease (PD-20% increase in lesion diameter), stable disease (SD-neither shrinkage nor increase of lesions).
Time Frame: 12 months
Population: Per Protocol Population
Measure: Number; unit: Percentage of Participants
Arm/Group | E7389 Intravenous 1.4 mg/m2
Number analyzed (Participants) | 105
Percentage of Participants
  Patients with measureable tumors | 59
  Complete Response | 0
  Partial Response | 8.1
  Stable Disease | 72.6
  Progressive Disease | 8.1
  Unknown | 11.3

ADVERSE EVENTS:
Arm/Group | E7389 Intravenous 1.4 mg/m2
Serious Adverse Events (participants affected / at risk) | 34/108
Other Adverse Events (participants affected / at risk) | 107/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E7389 Intravenous 1.4 mg/m2 (N=108)
Anemia (Blood and lymphatic system disorders) | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 2
Abdominal Pain (Blood and lymphatic system disorders) | 1
Diarrhea (Blood and lymphatic system disorders) | 2
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1
Melena (Gastrointestinal disorders) | 2
Esophageal Ulcer Hemorrhage (Gastrointestinal disorders) | 1
Chest Pain (General disorders) | 1
Edema Peripheral (General disorders) | 1
Pyrexia (General disorders) | 3
Suprpubic Pain (General disorders) | 1
Bradycardia (Cardiac disorders) | 2
Cardiac Arrest (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 2
Pharyngitis Streptococcal (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Sepsis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 2
Uriosepsis (Infections and infestations) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypovolemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Hemiparesis (Nervous system disorders) | 1
Spinal Cord Compression (Nervous system disorders) | 3
Confusional State (Psychiatric disorders) | 1
Bladder Obstruction (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Renal Colic (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 4
Renal Failure Acute (Renal and urinary disorders) | 1
Prostatic Pain (Reproductive system and breast disorders) | 1
Alveolitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3
Swelling Face (Skin and subcutaneous tissue disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Peripheral Ischemia (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E7389 Intravenous 1.4 mg/m2 (N=108)
Anemia (Blood and lymphatic system disorders) | 38
Leukopenia (Blood and lymphatic system disorders) | 30
Neutropenia (Blood and lymphatic system disorders) | 46
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Constipation (Gastrointestinal disorders) | 25
Diarrhea (Gastrointestinal disorders) | 28
Dry Mouth (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 26
Vomiting (Gastrointestinal disorders) | 11
Asthenia (General disorders) | 31
Fatigue (General disorders) | 47
Mucosal Inflammation (General disorders) | 6
Edema Peripheral (General disorders) | 19
Pain (General disorders) | 11
Pyrexia (General disorders) | 18
Urinary Tract Infection (Infections and infestations) | 10
Alanine Aminotransferase Increased (Investigations) | 7
Aspartate Aminotransferase Increased (Investigations) | 8
Anorexia (Metabolism and nutrition disorders) | 22
Dehydration (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 6
Underweight (Metabolism and nutrition disorders) | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Back Pain (Musculoskeletal and connective tissue disorders) | 11
Bone Pain (Musculoskeletal and connective tissue disorders) | 9
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 10
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 10
Dizziness (Nervous system disorders) | 8
Dysgeusia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 8
Neuropathy (Nervous system disorders) | 8
Neuropathy Peripheral (Nervous system disorders) | 15
Paraesthesia (Nervous system disorders) | 13
Insomnia (Psychiatric disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Alopecia (Skin and subcutaneous tissue disorders) | 20
Rash (Skin and subcutaneous tissue disorders) | 7
Hot Flush (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No